CLINICAL TRIAL: NCT02700711
Title: Randomized Clinical Trial: 03 (Methylphenidate and Duloxetine)
Brief Title: Methylphenidate-Duloxetine Combinations for Cocaine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Craig Rush, Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: RCT: 03; R56DA041201 (NIH)
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Methylphenidate; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo. Subjects will be maintained on placebo and methylphenidate during placebo maintenance.
  Interventions: Drug: Methylphenidate; Drug: Placebo
- Duloxetine (Experimental): Subjects will be maintained on oral duloxetine. Subjects will be maintained on placebo and methylphenidate during duloxetine maintenance.
  Interventions: Drug: Methylphenidate; Drug: Placebo; Drug: Duloxetine

INTERVENTIONS:
Drug: Methylphenidate — The pharmacodynamic effects of methylphenidate maintenance will be determined during maintenance on placebo and duloxetine.
  Other Names: Ritalin
Drug: Placebo — The pharmacodynamic effects of placebo will be determined during maintenance on placebo and duloxetine.
Drug: Duloxetine — The pharmacodynamic effects of duloxetine will be determined during maintenance on placebo and methylphenidate
  Other Names: Cymbalta
  Arms: Duloxetine

SUMMARY:
This study will determine the influence of methylphenidate (e.g., Ritalin®) and duloxetine (Cymbalta®), alone and in combination, on the cocaine use as measured by self-report and urine drug screens.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use
* Seeking treatment for cocaine use

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease or current unstable physical disease (e.g., past myocardial infarction, uncontrolled hypertension, diabetes, head trauma, seizures or CNS tumors) or current or past histories of serious psychiatric disorder or suicidal risk, other than substance abuse or dependence, will be excluded from research participation
* Females not currently using effective birth control
* Contraindications to cocaine, methylphenidate or duloxetine
* Currently using opioids for pain or who are currently maintained on methadone or buprenorphine for opioid use disorder will be excluded from participation
* Body weight less than 50 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Number of Cocaine Positive Urines | Six weeks
  Cocaine use will be assessed using qualitative urine drug screens over a six week period.

SECONDARY OUTCOMES:
Self-Reported Cocaine Use | Six weeks
  Cocaine use will be assessed using self-report on the Time Line Follow Back over a six week period.
Blood Pressure | Six weeks
  Blood Pressure in mmHG will be measured on each week day over a six week period.
Heart Rate | Six weeks
  Heart Rate in beats per minute will be measured on each week day over a six week period.
Side effects | Six weeks
  Subjects will complete a side effects questionnaire on each week day over a six week period. Side Effects questions will query subjects about common effects of centrally active medications.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared per NIH policy. Individual participant data will not be shared.